CLINICAL TRIAL: NCT01404676
Title: The Effect of Vildagliptin Based Treatment Versus Sulfonylurea on Glycemic Variability, Oxidative Stress, GLP-1, and Endothelial Function in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-02-053
Record Dates: First submitted 2010-06-22; First posted 2011-07-28 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Glucose variability; Oxidative stress; Endothelial cell function
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vildagliptin + Metformin (Experimental): Adding Vildagliptin to metformin users
  Interventions: Drug: Add Vildagliptin
- Glimepiride + Metformin (Active Comparator): Adding Glimepiride to metformin users
  Interventions: Drug: Add Glimepiride

INTERVENTIONS:
Drug: Add Vildagliptin — Adding Vildagliptin 50 mg bid to patients with type 2 diabetes mellitus being treated with metformin 500-1000mg bid per day who had hemoglobin A1c of 7.0-10.0%
  Arms: Vildagliptin + Metformin
Drug: Add Glimepiride — Adding Glimepiride 2mg to patients with type 2 diabetes mellitus being treated with metformin 500-1000mg bid per day who had hemoglobin A1c of 7.0-10.0%
  Arms: Glimepiride + Metformin

SUMMARY:
The effect of vildagliptin based treatment versus sulfonylurea based treatment on glycemic variability, oxidative stress, and endothelial function in patients with type 2 diabetes.

DETAILED DESCRIPTION:
Recently, improved understanding of the incretin effect on the pathophysiology of type 2 diabetes has led to development of new agent for hypoglycemic therapy. Vildagliptin is a potent and highly selective dipeptidyl peptidase-4 (DPP-4) inhibitor that augments the active glucagon-like peptide(GLP)-1 concentration, increases insulin secretion and improves glucose tolerance. Vildagliptin has a similar glucose lowering effect, but lower hypoglycemic events, as compared to glimepiride. Vildagliptin could improve not only the mean glycemic control but also 24 hour glycemic fluctuation by restoring the physiologic pattern of insulin and glucagon secretion. Furthermore, decreased postprandial glycemic excursion might reduce the oxidative stress markers and improve endothelial dysfunction. Those effects might be amplified in Asian patients because of prominent early phase insulin secretory defects accompanied with relatively less degree of insulin resistance. In addition, GLP-1 and GLP-1 analogues exert direct beneficial effects on endothelium-dependent vasodilatation. Therefore DPP-4 inhibitors may directly improve endothelial dysfunction.

Based on this assumption, this research will focus on the effect of vildagliptin on glycemic variability, oxidative stress markers and endothelial cell function compared to long acting sulfonylurea glimepiride in type 2 diabetic patients with inadequate glycemic control on metformin.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients with hemoglobin A1c levels within the range 7% - 10%

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change in mean amplitude of glycemic excursion(MAGE) for 12 weeks(12weeks - 0 week). | 0 week and 12 weeks
  To compare the effect of vildagliptin based treatment for 12 weeks on glycemic variability with sulfonylurea using continuous glucose monitoring system(CGMS).

SECONDARY OUTCOMES:
Change from baseline in oxidative stress markers and inflammatory markers at 12 weeks. Change from baseline in endothelial cell function at 12 weeks. | 0 week and 12 weeks
  1. To evaluate the change of oxidative stress markers and inflammatory markers from baseline.
  2. To evaluate the change of endothelial cell function using high-resolution ultrasonography to measure brachial artery flow-mediated dilation (FMD) from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Moon-Kyu Lee, Principal Investigator — Department of Internal Medicine, Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (1):
- Division of Endocrinology and Metabolism, Department of Internal Medicine, Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim G, Oh S, Jin SM, Hur KY, Kim JH, Lee MK. The efficacy and safety of adding either vildagliptin or glimepiride to ongoing metformin therapy in patients with type 2 diabetes mellitus. Expert Opin Pharmacother. 2017 Aug;18(12):1179-1186. doi: 10.1080/14656566.2017.1353080. Epub 2017 Jul 17. PMID 28714741